CLINICAL TRIAL: NCT00643175
Title: Effectiveness of Automated Inpatient Endocrinology Consultation for Osteoporotic Hip Fracture
Status: Terminated | Type: Observational
Why Stopped: Dr. Grose has left this practice, this study is terminated
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Andrew Grose, MD, SUNY Upstate Medical University
Other Study IDs: osteoporotic hip fracture
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Last update posted 2009-12-30 (Estimated); Status verified 2009-12

CONDITIONS: Osteoporosis
Keywords: The main objective is to have an endocrinologist treat osteoporosis in patients with fragility hip fractures.
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Osteoporosis in patients with fragility hip fractures.
  Interventions: Behavioral: Automated follow up

INTERVENTIONS:
Behavioral: Automated follow up — Treatment of osteoporosis after hip fracture is also being targeted as a future hospital quality assessment measure. Hospitals which have no plan in place to address osteoporosis treatment after hip fracture may be cited, and may have medicare money withheld. The goal of the study is to create an automated in-patient endocrinology consultation for osteoporotic hip fractures. We plan to gather patient data in a prospective manner including the endocrinologist recommendations, adherence to medical therapy after discharge, and future fracture rates. Planned interventions include only appropriate medical therapy for osteoporosis, DEXA bone scanning, and regularly scheduled telephone follow-up.

SUMMARY:
Osteoporosis has been called a "silent epidemic" whose prevalence is increasing. It often presents as a fragility fracture, with hospitalizations resulting from minimally traumatic hip fractures. While the fractures are treated appropriately, the underlying pathology is often ignored. Numerous studies have shown that prior fracture increases the risk for further fracture. In 2004 the Surgeon General released a report on osteoporosis, the details of which include multi-disciplinary treatment of osteoporotic fractures. Treatment of osteoporosis after hip fracture is also being targeted as a future hospital quality assessment measure. Hospitals which have no plan in place to address osteoporosis treatment after hip fracture may be cited, and may have medicare money withheld. The goal of the study is to create an automated in-patient endocrinology consultation for osteoporotic hip fractures. We plan to gather patient data in a prospective manner including the endocrinologist recommendations, adherence to medical therapy after discharge, and future fracture rates. Possible planned interventions include only appropriate medical therapy for osteoporosis, DEXA bone scanning, and regularly scheduled telephone follow-up.

ELIGIBILITY:
Inclusion:

1. over 55
2. non-traumatic hip fracture

Exclusion criteria:

1. currently on anti-osteoporosis pharmacotherapy including bisphosphonates, PTH, and calcitonin
2. high energy nature of fracture, including MVA, fall from height greater than 3 feet
3. severe dementia, lack of capacity

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Using the existing WebCAIS order system, an automated endocrinology consult and appropriate laboratory studies will be drawn on all non-traumatic hip fractures. Data from these patients will be collected in a prospective study, and the patients will be followed up over time to check adherence to osteoporotic medical therapy and future incidence of re-fracture.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2007-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States